CLINICAL TRIAL: NCT02856217
Title: Comparison of the Tunneling or Non-tunneling During Minimally Invasive Sacrocolpopexy in Terms of Lower Urinary Tract and Bowel Symptoms.
Brief Title: Impact of Tunneling During Minimally Invasive Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-0157
Record Dates: First submitted 2016-07-25; First posted 2016-08-04 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Lower Urinary Tract Symptoms; Lower Gastrointestinal Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tunneling (Active Comparator): Placement of mesh between vaginal apex and sacrum is retroperitoneally placed in peritoneal tunneling in SCP: creating a tunnel between vaginal apex and sacrum under peritoneum without disturbing the integrity of the peritoneum.
  Interventions: Procedure: tunneling
- non-tunneling (Active Comparator): Placement of mesh between vaginal apex and sacrum is retroperitoneally placed in peritoneal non-tunneling group in SCP: incised and sutured peritoneum between vaginal apex and sacrum
  Interventions: Procedure: non-tunneling

INTERVENTIONS:
Procedure: tunneling — In this arm of the study which is Peritoneal tunneling group in SCP, standard minimal invasive sacrocolpopexy procedure will be performed. Placement of mesh between vaginal apex and sacrum is retroperitoneally (creating a tunnel between vaginal apex and sacrum under peritoneum without disturbing the integrity of the peritoneum)
  Other Names: Peritoneal tunneling during minimal invasive sacrocolpopexy
  Arms: tunneling
Procedure: non-tunneling — In this arm of the study which is Peritoneal non-tunneling group in SCP, standard minimal invasive sacrocolpopexy procedure will be performed. Placement of mesh between vaginal apex and sacrum is retroperitoneally (incised and sutured peritoneum between vaginal apex and sacrum).
  Other Names: Peritoneal non-tunneling during minimal invasive SCP
  Arms: non-tunneling

SUMMARY:
Pelvic organ prolapse occurs when the uterus or vaginal walls bulge into or beyond the vaginal introitus. Abdominal sacrocolpopexy is the most durable operation for advanced pelvic organ prolapse and serves as the criterion standard against which other operations are compared. Abdominal sacrocolpopexy involves attaching the vaginal apex to the sacral anterior longitudinal ligament reinforced with a graft, usually synthetic mesh. More than 225.000 surgeries are performed annually in the United States for pelvic organ prolapse. Abdominal sacrocolpopexy is considered the most durable pelvic organ prolapse surgery, but little is known about safety and long-term effectiveness.

Purpose of this study is to compare effect of tunneling or non-tunneling mesh placement on lower urinary tract symptoms and bowel symptoms in patients who underwent surgery with laparoscopic or robot-assisted sacrocolpopexy which is accepted surgical procedures for pelvic organ prolapse.

DETAILED DESCRIPTION:
Pelvic organ prolapse represents a common female pelvic floor disorder that increases with age and has a serious impact on quality of life. It is estimated that 30% of women aged 50-89 years will seek consultation for pelvic floor disorders. The purpose of any surgical repair of pelvic organ prolapse is to restore pelvic anatomy, preserving urinary, intestinal, and sexual function, with the lowest rate of recurrences and complications.

In the history of surgical repair for pelvic organ prolapse vaginal or abdominal approach has been performed. In spite of decreased morbidity and shorter hospitalisation advantage with vaginal procedures, they have consistently lower long-term success rates compared to abdominal sacrocolpopexy. In contrast, the abdominal approach is considered the gold standard for surgical correction of vaginal vault prolapse, with reported long-term efficacy rates. However, the associated morbidity of open laparotomy has made this procedure less favourable. In an effort to overcome these drawbacks, a minimally invasive laparoscopic approach has been adopted. However, the rigidity of the laparoscopic instrumentation makes intracorporeal suturing and dissection in the narrow pelvis challenging. Robot-assisted technology, with its stereoscopic vision and the use of instruments which easily moved by wrist movement, offers an ergonomic platform that simplifies complex laparoscopic tasks and has been widely adopted by pelvic surgeons.

Most complications following sacrocolpopexy can occur with either an open or a minimally invasive approach, typically at similar rates. Bladder injury, postoperative voiding dysfunction and lower urinary tract symptoms may occur. Lower urinary tract symptoms may develop postoperatively for reason that are still not clearly understood. De nova lower urinary tract symptoms may appear after laparoscopic or robot-assisted sacrocolpopexy with a range from 0% to 27%. As with urinary system complication, bowel complications (bowel injury, bowel dysfunction) may occur intraoperatively and postoperatively. Constipation is the mostly reported with a range from 0% to 19%. Retroperitonealization of the mesh used in laparoscopic sacrocolpopexy or robot-assisted sacrocolpopexy is thought to reduce the risk of bowel injury, although some authors have noted a lack of bowel injuries when the mesh was left exposed to the peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is at least 18 years of age
* Subject is who can English speaking and reading
* Subject must have documented diagnosis of apical vaginal prolapse with leading edge of pelvic organ prolapse at or beyond the hymen. At or beyond the hymen is defined as Pelvic Organ Prolapse Quantification System (POP-Q) scores of C ≥ -1/2 total vaginal length (TVL)
* Subject reports a bothersome bulge they can see or feel per Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20), question 3, response of 2 or higher (i.e., responses of "somewhat", "moderately", or "quite a bit")
* Subject or subject's legally authorized representative is willing to provide written informed consent
* Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

* Subject is pregnant or intends to become pregnant during the study
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI) or tissue necrosis
* Subject has history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Subject has systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan's syndrome, Ehlers Danlos, collagenosis, polymyositis or polymyalgia rheumatica)
* Subject has uncontrolled diabetes mellitus (DM)
* Subject has a known neurologic or medical condition affecting bladder function (e.g., multiple sclerosis, spinal cord injury or stroke with residual neurologic deficit)
* Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
* Subject is currently participating in or plans to participate in another device or drug study during this study
* Subject has a known sensitivity to polypropylene
* Subject has had previous prolapse repair with mesh (abdominal or vaginal)
* Subject is planning to undergo a concomitant vaginal repair with use of mesh

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Lower Urinary Tract Symptoms | Up to 1 year
  In follow-up, using questionnaires specifically, Pelvic Floor Distress Inventory Questionnaire - Short Form 20 will be used in preoperatively, in 2.week visit, 6.week visit and 12.months visit.

SECONDARY OUTCOMES:
Pelvic Organ Prolapse | Up to 1 year
  In follow-up, using questionnaires specifically, Pelvic Floor Distress Inventory Questionnaire - Short Form 20 will be used in preoperatively, in 2.week visit, 6.week visit and 12.months visit.
Lower Gastrointestinal Tract Symptoms | Up to 1 year
  In follow-up, using questionnaires specifically, Pelvic Floor Distress Inventory Questionnaire - Short Form 20 will be used in preoperatively, in 2.week visit, 6.week visit and 12.months visit.
Surgical duration (time from skin incision to skin closure) | Postoperative 1.day
  Outcome will be collected from patients operation files
Blood loss | Postoperative 1.day
  Outcome will be collected from patients operation files and anesthesiology notes
Intraoperative complications (conversion to open procedure or inadvertent structural lesions such as bladder, bowel, vessels, or solid organs) | Postoperative 1.day
  Outcome will be collected from patients operation files and prospectively will be noted from surgeon who is the PI of the study.
Postoperative complications (Clavien-Dindo classification) | Postoperative 7.day
  The Clavien-Dindo Classification of Surgical Complications questionnaires will be used to collect the complications
Sexual function | Up to 1 year
  Evaluation of patient's sexual function with Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan S Kilic, MD, Principal Investigator — UTMB, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maher C, Feiner B, Baessler K, Glazener CM. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD004014. doi: 10.1002/14651858.CD004014.pub4. PMID 20393938
- [Result] Luber KM, Boero S, Choe JY. The demographics of pelvic floor disorders: current observations and future projections. Am J Obstet Gynecol. 2001 Jun;184(7):1496-501; discussion 1501-3. doi: 10.1067/mob.2001.114868. PMID 11408873
- [Result] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Result] Karram M, Goldwasser S, Kleeman S, Steele A, Vassallo B, Walsh P. High uterosacral vaginal vault suspension with fascial reconstruction for vaginal repair of enterocele and vaginal vault prolapse. Am J Obstet Gynecol. 2001 Dec;185(6):1339-42; discussion 1342-3. doi: 10.1067/mob.2001.119077. PMID 11744906
- [Result] Benson JT, Lucente V, McClellan E. Vaginal versus abdominal reconstructive surgery for the treatment of pelvic support defects: a prospective randomized study with long-term outcome evaluation. Am J Obstet Gynecol. 1996 Dec;175(6):1418-21; discussion 1421-2. doi: 10.1016/s0002-9378(96)70084-4. PMID 8987919
- [Result] Nygaard IE, McCreery R, Brubaker L, Connolly A, Cundiff G, Weber AM, Zyczynski H; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy: a comprehensive review. Obstet Gynecol. 2004 Oct;104(4):805-23. doi: 10.1097/01.AOG.0000139514.90897.07. PMID 15458906
- [Result] Ganatra AM, Rozet F, Sanchez-Salas R, Barret E, Galiano M, Cathelineau X, Vallancien G. The current status of laparoscopic sacrocolpopexy: a review. Eur Urol. 2009 May;55(5):1089-103. doi: 10.1016/j.eururo.2009.01.048. Epub 2009 Feb 4. PMID 19201521
- [Result] Rosenblum N. Robotic approaches to prolapse surgery. Curr Opin Urol. 2012 Jul;22(4):292-6. doi: 10.1097/MOU.0b013e328354809c. PMID 22647648
- [Result] Lee RK, Mottrie A, Payne CK, Waltregny D. A review of the current status of laparoscopic and robot-assisted sacrocolpopexy for pelvic organ prolapse. Eur Urol. 2014 Jun;65(6):1128-37. doi: 10.1016/j.eururo.2013.12.064. Epub 2014 Jan 8. PMID 24433811
- [Result] Gadonneix P, Ercoli A, Salet-Lizee D, Cotelle O, Bolner B, Van Den Akker M, Villet R. Laparoscopic sacrocolpopexy with two separate meshes along the anterior and posterior vaginal walls for multicompartment pelvic organ prolapse. J Am Assoc Gynecol Laparosc. 2004 Feb;11(1):29-35. doi: 10.1016/s1074-3804(05)60006-0. PMID 15104827